CLINICAL TRIAL: NCT06166667
Title: Effect of Fecal Capsule on Chronic Kidney Disease (CKD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Provincial People's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: (2022) SYKLSZ No.352
Record Dates: First submitted 2023-05-06; First posted 2023-12-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental): Fecal Microbiota Transplant
  Interventions: Procedure: Fecal Microbiota Transplant（FMT）

INTERVENTIONS:
Procedure: Fecal Microbiota Transplant（FMT） — Patients involved in the trial received 20 capsules of Enterobacteriaceae (one course) on days 1, 8, and 15, which were provided by Dongyuan Yikang company. Patients were prohibited from taking antibiotics such as amoxicillin and Cefalexin during the trial.

SUMMARY:
By collecting blood, urine and stool samples before and after oral Enterobacteriaceae capsule (FMT) from CKD subjects, we investigated the role and related mechanisms of gut microecology in the development of CKD using a combination of metagenomic sequencing, metabolomic analysis and flow cytometry.

DETAILED DESCRIPTION:
Patients involved in the trial received 16 capsules of Enterobacteriaceae (one course) on days 1, 8, and 15, which were provided by Dongyuan Yikang company. Patients were prohibited from taking antibiotics such as amoxicillin and Cefalexin during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects: Patients with chronic kidney disease (CKD)
2. GFR ≥ 30 ml / min, or serum creatinine ≤ 442 μ mol/L
3. Negative urine pregnancy test and no plans for pregnancy for the next 18 months, enabling effective contraception
4. Age: 18-70 years
5. Signed informed consent for clinical studies informed consent for treatment of patients with flora transplantation (FMT)

Exclusion Criteria:

1. Had taken antibiotics for nearly 14 days
2. Active systemic infections or severe infections within 1 month prior to enrollment, including HIV, HBV, HCV
3. White blood cell count < 3.0x109/l; Platelet count < 80x109 / L, or had other hematologic diseases
4. Presence of malignancy and other diseases with expected survival time < 3 months
5. Presence of IBD, CDI, or gastrointestinal tumors
6. Presence of active gastrointestinal bleeding or acute and chronic gastrointestinal inflammation
7. Were or had undergone FMT
8. Psychosis and cognitive impairment
9. History of alcohol or drug abuse
10. Pregnant or lactating women
11. Difficult to follow-up
12. Difficult or unwilling to cooperate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Abundance of gut microbiota | 6 months after the end of the trial
  Fecal sample metagenomic sequencing

SECONDARY OUTCOMES:
24-hour urine protein quantitative change rate | 6 months after the end of the trial
  Urine sample
the density of immune cells | 6 months after the end of the trial
  Blood samples
Cytokine concentration | 6 months after the end of the trial
  Blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Yafeng Li, Professor, Principal Investigator — Shanxi Provincial People's Hospital (Fifth Hospital) of Shanxi Medical University
Locations (1):
- Shanxi Provincial People's Hospita, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed，ResMan,http://www.medresman.org.cn
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the study is completed
Access Criteria: Nephrologist